CLINICAL TRIAL: NCT04645264
Title: Effect of Indwelling Foley Placement, Immediate Post-Operative Straight Catheterization, or No Catheterization on Post-operative Urinary Retention After Transforaminal Lumbar Interbody Fusions
Brief Title: Effect of Catheter on Postoperative Urinary Retention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI initiated closure due to limited clinical resources and lack of participation.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Research Manger, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18080302
Record Dates: First submitted 2019-09-06; First posted 2020-11-27 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Transforaminal Lumbar Interbody Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Indwelling Foley (Experimental): Indwelling Foley placed during surgery
  Interventions: Device: Foley Catheter
- Straight Catheter (Active Comparator): straight catheterization (in-and-out straight catheterization) will take place at the end of the surgery
  Interventions: Device: Foley Catheter
- No Catheter (No Intervention): Patient is not catheterized

INTERVENTIONS:
Device: Foley Catheter — The patient is catheterized during surgery.
  Arms: Indwelling Foley; Straight Catheter

SUMMARY:
To determine if indwelling Foley placement at the onset of the procedure, straight catherization at the conclusion of the procedure, or no catheterization produces the lowest rates of postoperative urinary retention after transforaminal lumbar interbody fusions (TLIFs).

DETAILED DESCRIPTION:
Post-operative urinary retention (POUR) is one the most common post-operative complications after elective spine surgeries. Common causes of postoperative urinary retention (POUR) include bladder stenosis, distension, trauma due to catheterizations, age, and prostate hyperplasia. The incidence of POUR increases with age, gender, types of surgery conducted, any comorbidities such as cerebral palsy or multiple sclerosis, use of drugs such as anticholinergic agents, beta blockers, or sympathomimetics, and use of IV fluids.

This condition has been associated with the development of UTIs and sepsis, increased post-operative length of stay (LOS), and 90-day readmission after surgery. In the field of spine surgery, the reported incidence of POUR is highly variable, and there is no consensus on effective methods of prevention. We set out to assess POUR from patients catheterized compared to non-catheterized following a transforaminal lumbar interbody fusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary single-level MIS TLIF (Diagnosis: radiculopathy, stenosis, herniated nucleus pulposus, degenerative disc disease, spondylosis, osteophytic complexes, spondylolysis, spondylolisthesis)
* Patients able to provide informed consent

Exclusion Criteria:

* Patients with baseline urinary dysfunction requiring manual bladder emptying via intermittent straight catheterization, suprapubic catheters, or other indwelling catheters. -Allergies or other contraindications to medicines in the post- operative urinary retention protocol
* Lack of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indwelling Foley | Straight Catheter | No Catheter
Started | 3 | 2 | 2
Completed | 3 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indwelling Foley | Straight Catheter | No Catheter | Total
Number analyzed (Participants) | 3 | 2 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 55 [46 to 60] | 57 [55 to 58] | 58 [55 to 66] | 57 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 1 | 1 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: How long was the patients post-operative stay?
Time Frame: Date of surgery until the date of hospital discharge, up to 1 month
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Indwelling Foley | Straight Catheter | No Catheter
Number analyzed (Participants) | 3 | 2 | 2
days | 3 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: From the date of surgery to 6 months post-surgical
Arm/Group | Indwelling Foley | Straight Catheter | No Catheter
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04645264/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04645264/ICF_002.pdf